CLINICAL TRIAL: NCT01011751
Title: Efficacy and Tolerance of Cyproterone Acetate Versus Medroxyprogesterone Acetate Versus Venlafaxine LP in the Treatment of Hot Flushes Caused by Leuprorelin 11.25 mg in Patients Treated for a Prostate Adenocarcinoma
Brief Title: Treatment of Hot Flushes Caused by Leuprorelin 11.25 mg in Prostate Adenocarcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F-LEU-100; U1111-1169-6822 (Registry Identifier: WHO)
Record Dates: First submitted 2009-11-03; First posted 2009-11-11 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Adenocarcinoma, Prostate
Keywords: Drug Therapy
MeSH Terms: conditions — Adenocarcinoma | interventions — Cyproterone Acetate; Medroxyprogesterone Acetate; Venlafaxine Hydrochloride; Leuprolide; Flutamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cyproterone acetate (Experimental): Leuprorelin 11.25 mg, injection, subcutaneously at Months 0, 3, and 6, and flutamide 250 mg, tablet, orally, thrice daily for first 30 days from first leuprorelin administration. From Month 6, cyproterone acetate 50 mg, tablet-in-capsule, along with cyproterone acetate placebo-matching capsule, orally, once daily in the morning and cyproterone acetate 50 mg, tablet-in-capsule, orally, once daily in the evening for 8 weeks. Cyproterone acetate placebo-matching capsule, orally, once daily in the morning for the next 2 weeks.
  Interventions: Drug: Cyproterone acetate; Drug: Leuprorelin; Drug: Flutamide; Drug: Placebo
- Medroxyprogesterone acetate (Experimental): Leuprorelin 11.25 mg, injection, subcutaneously at Months 0, 3, and 6, and flutamide 250 mg, tablet, orally, thrice daily for first 30 days from first leuprorelin administration. From Month 6, medroxyprogesterone acetate 10 mg, tablet-in-capsule, along with medroxyprogesterone acetate placebo-matching capsule, orally, once daily in the morning and medroxyprogesterone acetate 10 mg, tablet-in-capsule, orally, once daily in the evening for 8 weeks. Medroxyprogesterone acetate placebo-matching capsule, orally, once daily in the morning for the next 2 weeks.
  Interventions: Drug: Medroxyprogesterone acetate; Drug: Leuprorelin; Drug: Flutamide; Drug: Placebo
- Venlafaxine (Experimental): Leuprorelin 11.25 mg, injection, subcutaneously at Months 0, 3, and 6, and flutamide 250 mg, tablet, orally, thrice daily for first 30 days from first leuprorelin administration. From Month 6, venlafaxine 75 mg, capsule, orally, once daily in the morning and venlafaxine placebo-matching capsule, orally, once daily in the evening for 8 weeks. Venlafaxine 37.5 mg, capsule, orally, once daily in the evening for the next 2 weeks.
  Interventions: Drug: Venlafaxine; Drug: Leuprorelin; Drug: Flutamide; Drug: Placebo

INTERVENTIONS:
Drug: Cyproterone acetate — Cyproterone acetate tablet-in-capsule.
  Other Names: Androcur® 50 mg
  Arms: Cyproterone acetate
Drug: Medroxyprogesterone acetate — Medroxyprogesterone acetate tablet-in-capsule.
  Other Names: Gestoral® 10 mg
  Arms: Medroxyprogesterone acetate
Drug: Venlafaxine — Venlafaxine capsule.
  Other Names: Effexor® LP 37.5 mg
  Arms: Venlafaxine
Drug: Leuprorelin — Leuprorelin injection.
  Other Names: Enantone® 11.25 mg
Drug: Flutamide — Flutamide tablet
Drug: Placebo — Cyproterone acetate, medroxyprogesterone acetate or venlafaxine placebo-matching capsule.

SUMMARY:
The purpose of this study is to compare the efficacy of three drugs (cyproterone acetate, medroxyprogesterone acetate and venlafaxine) in the treatment of hot flushes caused by leuprorelin LP 11.25 milligram (mg) in participants suffering from prostate cancer.

DETAILED DESCRIPTION:
Three drugs will be tested in this study: cyproterone acetate, medroxyprogesterone acetate and venlafaxine. Cyproterone acetate, medroxyprogesterone acetate and venlafaxine are being tested to treat men who suffer from hot flushes due to androgen suppression treatment for prostate cancer. This study will look at the frequency and severity of hot flushes caused by leuprorelin in participants who will take cyproterone acetate, medroxyprogesterone acetate or venlafaxine. The study will randomize approximately 311 participants. All participants will receive 2 injections of leuprorelin 11.35 mg at Months 0 and 3 along with flutamide tablets in the first month of treatment to prevent flare-up. After 6 months, eligible participants will receive third injection of leuprorelin and will be randomly assigned to one of the three treatment groups-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Cyproterone acetate (Androcur® 50 mg)
* Medroxyprogesterone acetate (Gestoral® 10 mg)
* Venlafaxine (Effexor® LP 37.5 mg) All participants will be asked to take 2 capsules in the morning and 1 capsule in the evening for 10 weeks. All participants will be asked to complete the self-evaluation hot-flushes (HF) questionnaire daily for 12 weeks from the start of treatment for hot flushes.

This multi-center trial will be conducted in France. The overall time to participate in this study is approximately 9 months. Participants will make 5 visits to the clinic during the study.

ELIGIBILITY:
Inclusion Criteria: - Patient has a histologically proven prostatic adenocarcinoma.

* Patient has been on a gonadotropin releasing hormone (GnRH) agonist treatment for a duration of at least 1 year.
* Karnofsky index greater than or equal to (>=) 70 %.
* Patient who, after having been clearly informed, has given his written consent to participate in the study.

Exclusion Criteria:

* Patient included in a therapeutic trial in the 3 months preceding the inclusion visit.
* Prescription of agonist planned in the context of neo-adjuvant hormonotherapy.
* Patient has symptomatic bone metastases.
* Patient already treated with hormonotherapy for his prostate cancer or has received a hormonal treatment other than a GnRH agonist for this cancer (apart from palliative care of flare-up with anti-androgens).
* Patient is unable to understand the information regarding the study provided to him, of giving his consent or who has refused to sign the informed consent sheet.
* Patient for whom risk follow up could not be guaranteed within the conditions stipulated in the protocol or is unable to complete the self-evaluation questionnaires.
* Diabetic, or patient with severe progressive disease: kidney, liver, cardiovascular (especially high uncontrolled BP), psychiatric.
* Has a Thromboembolic history or concomitant thromboembolic disease.
* Patient had hepatocellular insufficiency or hepatic cytolysis (serum glutamic oxaloacetic transaminase / serum glutamic pyruvate transaminase [SGOT/SGPT] >3 times laboratory normal range).
* Patient had a contra-indication to one of the study drugs.
* Patient receiving corticotherapy or concomitant prescription for non-selective monoamine oxidase inhibitors (MAOI), serotonin re-uptake inhibitors, clonidine, gabapentine, veripride, tibolone or beta-alanine.
* Patient was undergoing medical treatment for a depressive phase or had been treated for this during the previous 2 years before inclusion.
* Patient with a history of congenital galactosemy, poor absorption of glucose or galactose syndrome or even a lactase deficiency.
* Patient had another cancer in the 5 previous years excluding basocellular epithelioma or in situ carcinoma.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2004-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Percent Change from Randomization in Hot Flushes (HF) Score at Week 4 of Treatment | Randomization (Month 6) and Week 4 of treatment (Month 7)
  The change is calculated as follows: [(HF score at Week 4 of treatment - HF score at randomization)/HF score at randomization]*100. The calculation of the HF score will be done as follows: a coefficient is allocated to each severity grade, it varies from 1 to 4 (1: slight; 2: moderate; 3: severe; 4: very severe), and the calculation of the daily score is equal to the sum of the daily instances of hot flushes multiplied by their severity coefficient. The score calculated at randomization and Week 4 of treatment will be the average of the scores recorded in the preceding week. The score range will depend upon the frequency of hot flushes, and higher score signifies higher severity of hot flushes.

SECONDARY OUTCOMES:
Percent Change from Randomization in HF Frequency at Weeks 4, 8 of Treatment and Last Available Value | Randomization (Month 6), Weeks 4 and 8 of treatment (Months 7 and 8, respectively) and last available value (Month 7 or 8)
  The change is calculated as follows: [(HF frequency at specified Week of treatment - HF frequency at randomization)/HF score at randomization]*100.
Percentage of Participants With More Than 50 percent (%) Decrease in HF Score | Week 4 of treatment
  The percentage of participants with at least 50 % improvement in HF score after 4 weeks of treatment compared to randomization will be calculated. The calculation of the HF score will be done as follows: a coefficient is allocated to each severity grade, it varies from 1 to 4 (1: slight; 2: moderate; 3: severe; 4: very severe), and the calculation of the daily score is equal to the sum of the daily instances of hot flushes multiplied by their severity coefficient. The score range will depend upon the frequency of hot flushes, and higher score signifies higher severity of hot flushes. The score calculated at randomization and Week 4 of treatment will be the average of the scores recorded in the preceding week.
Percentage of Participants with Complete Regression of hot flushes | Week 4 of treatment
  Complete regression at Week 4 of treatment signifies complete disappearance of hot flushes upon 4 weeks of treatment.
Percentage of Participants With A Decrease in the Level of HF Complaint | Weeks 4 and 8 of treatment and Week 12 after the start of treatment
  Decrease (improvement) in the level of complaint regarding hot flushes will be assessed compared to randomization. Participants' level of complaints about hot flushes was recorded at each visit of the study. The change in the level of complaints will be classified as degradation, non-change or improvement.
Percent Change in HF Score from Randomization at Week 8 of Treatment and Last Available Value | Randomization, Week 8 of treatment, and last available value (Month 7 or 8)
  The change is calculated as follows: [(HF score at specified Week of treatment - HF score at randomization)/HF score at randomization]*100. The calculation of the HF score will be done as follows: a coefficient is allocated to each severity grade, it varies from 1 to 4 (1: slight; 2: moderate; 3: severe; 4: very severe), and the calculation of the daily score is equal to the sum of the daily instances of hot flushes multiplied by their severity coefficient. The score range will depend upon the frequency of hot flushes, and higher score signifies higher severity of hot flushes. The score calculated at randomization and Week 8 of treatment will be the average of the scores recorded in the preceding week.
Percent Change from Week 4 of treatment in HF Score at Week 8 of Treatment | Weeks 4 and 8 of treatment
  The change is calculated as follows: [(HF score at Week 8 of treatment - HF score at Week 4 of treatment)/HF score at Week 4 of treatment]*100. The calculation of the HF score will be done as follows: a coefficient is allocated to each severity grade, it varies from 1 to 4 (1: slight; 2: moderate; 3: severe; 4: very severe), and the calculation of the daily score is equal to the sum of the daily instances of hot flushes multiplied by their severity coefficient. The score range will depend upon the frequency of hot flushes, and higher score signifies higher severity of hot flushes. The score calculated at Weeks 4 and 8 of treatment will be the average of the scores recorded in the preceding week.
Percent Change from Week 4 of treatment in HF Frequency at Week 8 of Treatment | Weeks 4 and 8 of treatment
  The change is calculated as follows: [(HF frequency at Week 8 of treatment - HF frequency at Week 4 of treatment)/HF score at Week 4 of treatment]*100.
Percentage of Participants Who Wish to Continue the Treatment at the End of Week 10 | Weeks 8 and 12 after the start of treatment
  Participants will be asked at Week 8 and 12 visits if they would like to continue the study treatment beyond the protocol-specified 10 weeks of treatment.
Percentage of Participants Who Wish to Restart the Treatment at the End of Week 12 | Week 12 after the start of treatment
  Participants will be asked at Week 12 visit if they would like to restart the study treatment which ended after 10 weeks.
European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (EORTC QLQ-C30) | Baseline (Month 0), randomization (Month 6), Weeks 4 and 8 of treatment, Week 12 after the start of treatment
  EORTC QLQ-C30: includes functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). Most questions uses 4 point scale (1 'Not at all' to 4 'Very much'; 2 questions uses 7-point scale (1 'very poor' to 7 'Excellent'). Scores are averaged and transformed to 0-100 scale; for the 5 functional scales and the global quality-of-life scale, a higher score represents a better level of functioning. For the symptom-oriented scales and items, a higher score corresponds to a higher level of symptoms.
Participant's Satisfaction About Treatment | Week 4, 8 of treatment, and Week 12 after the start of treatment
  Participant's satisfaction is assessed by asking them how they would rate the treatment efficacy as not very effective, moderately effective and very effective at 4, 8 weeks of treatment and 12 weeks after the start of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: jacques irani, MD, Principal Investigator — Poitiers hospital
Locations (1):
- Professor Jacques IRANI, Poitiers, Poitiers, France

REFERENCES:
- [Derived] Irani J, Salomon L, Oba R, Bouchard P, Mottet N. Efficacy of venlafaxine, medroxyprogesterone acetate, and cyproterone acetate for the treatment of vasomotor hot flushes in men taking gonadotropin-releasing hormone analogues for prostate cancer: a double-blind, randomised trial. Lancet Oncol. 2010 Feb;11(2):147-54. doi: 10.1016/S1470-2045(09)70338-9. Epub 2009 Dec 4. PMID 19963436